CLINICAL TRIAL: NCT05493215
Title: A Phase 2 Study of Imatinib Therapeutic Drug Monitoring in Gastrointestinal Stromal Tumor
Brief Title: Imatinib TDM in GIST
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Reema A. Patel (Other)
Responsible Party: Sponsor-Investigator, Reema A. Patel, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-23-GI-131
Record Dates: First submitted 2022-08-05; First posted 2022-08-09 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Gastrointestinal Stromal Tumors
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Imatinib TDM (Experimental): Patients with diagnosed gastrointestinal stromal tumor (GIST) who are currently being treated with imatinib.
  Interventions: Drug: Imatinib

INTERVENTIONS:
Drug: Imatinib — Therapeutic drug level monitoring with plans to increase to adjust drug dosage based on levels and patient symptoms.
  Other Names: Gleevec

SUMMARY:
Imatinib can lead to long recurrence free survival in patients diagnosed with gastrointestinal stromal tumors (GIST); however side effects can significantly hinder quality of life for our patients. This study will use therapeutic drug monitoring to improve quality of life and symptoms and assess how many patients maintain therapeutic levels. Free drug levels and pharmokinetics of imatinib will also be monitored.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed GIST with KIT mutation or PDGFRA mutation (non-D842V)
* Currently receiving imatinib initiated within the last 3 months or to be started in the next 1 month
* Prior systemic chemotherapy for other malignancy is allowed as long as it was completed within the past 6 months and there is no evidence of disease
* Age ≥18 years
* ECOG performance status of 0 or 1
* Normal organ function

Exclusion Criteria:

* Presence of PDGFRA D842V mutation
* Known allergy to imatinib or allergic reactions to compounds of similar chemical or biologic composition to the study drug
* Concomitant anticoagulation with oral warfarin.
* Use of strong inhibitors or inducers of CYP3A or CYP3A4, drugs metabolized by CYP3A4 or CYP2D6
* Uncontrolled intercurrent illness
* Concurrent malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2024-03-26 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Grade 3/4 adverse events attributable to imatinib per CTCAE v5.0 | 6 months
  To compare the incidence of Grade 3/4 adverse events attributable to imatinib per CTCAE v5.0 in patients who receive therapeutic drug monitoring (TDM) with imatinib to a historical control.

SECONDARY OUTCOMES:
Percent of patients achieving therapeutic levels of imatinib. | 6 months
  Percent of patients achieving therapeutic levels of imatinib.
Quality of Life based on the EORTC QLQ-C30 | 6 months
  Quality of Life will be assessed using the EORTC Core Quality of Life questionnaire (EORTC QLQ-C30). The EORTC QLQ-C30 is designed to measure cancer patients' physical, psychological and social functions. It incorporates five functional scales, three symptom scales, a global health status, financial impact, and single items assessing additional symptoms. All scales and single-item measures are transformed so that scores range from 0-100; higher scores represent a higher response level.
Average dose of imatinib required to achieve therapeutic levels and drug dose over 3 years | 3 year

CONTACTS AND LOCATIONS:
Overall Officials: Reema Patel, MD, Principal Investigator — University of Kentucky
Locations (1):
- Markey Cancer Center, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No